CLINICAL TRIAL: NCT03311464
Title: A Phase 3 Multicenter, Open-Label, Single Arm Study of the Efficacy and Safety of Adalimumab in Active Ulcer(s) of Pyoderma Gangrenosum in Subjects in Japan
Brief Title: A Study Assessing the Efficacy and Safety of Adalimumab in Active Ulcer(s) of Pyoderma Gangrenosum in Participants in Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M16-119
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Pyoderma Gangrenosum
Keywords: Pyoderma Gangrenosum; Ulcer; Efficacy; Safety; Adalimumab; Humira®; Japan
MeSH Terms: conditions — Pyoderma Gangrenosum; Ulcer | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm A (Experimental): Participants receiving adalimumab for Pyoderma Gangrenosum active ulcer(s).
  Interventions: Drug: adalimumab

INTERVENTIONS:
Drug: adalimumab — Study drug will be administered subcutaneously.
  Other Names: Humira®

SUMMARY:
This study is designed to investigate the efficacy, safety and pharmacokinetics of adalimumab in subjects in Japan with active ulcer(s) due to Pyoderma Gangrenosum (PG).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be able and willing to provide written informed consent. If the participant is < 20 years old, a parent or legal guardian must be willing to give written informed consent
* Participants must have a diagnosis of ulcerative (classic) PG made by the Investigator
* Participants must have demonstrated an inadequate response to conventional PG therapy or in the opinion of the Investigator they are not a suitable candidate for conventional PG treatment.

Exclusion Criteria:

* Participants with pustular, bullous/atypical, or vegetative variants of PG
* Participants with clinical evidence of ulceration that is non-PG related, vasculitis, thrombosisprone conditions, or monoclonal gammopathy
* Participants with a histopathological finding that is consistent with a diagnosis other than PG
* Participants receiving a therapeutic dose of prednisolone
* Participants with prior exposure to adalimumab or previous participation in an adalimumab clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2020-04-21 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who have achieved target Pyoderma Gangrenosum Area Reduction (PGAR) | Week 26
  The participants will be assessed whether they meet target PGAR at Week 26 based on PGAR score.

SECONDARY OUTCOMES:
Proportion of participants achieving Physician's Global Assessment (PGA) 0 or 1 | Week 6 and Week 26
  The Investigator assesses the global improvement of all ulcers including the target ulcer according to the scales at the specified visits.
Mean time to occurrence of new PG ulcers | Up to Week 26
  A new PG ulcer is defined as not present at Baseline and not caused by the epithelial bridging of an existing ulcer at Baseline. The time after Baseline when the new lesion was observed will be recorded.
Change from Baseline in total number of active ulcers | Week 26
  The number of all active PG ulcers will be counted at the specified visits.
Change from Baseline in Dermatology Life Quality Index (DLQI) | Week 6 and Week 26
  The DLQI will be used to assess the symptoms and the impact of skin problems on quality of life.
Changes from Baseline in total ulcer area | Week 6 and Week 26
  The change in total ulcer area is assessed.
Proportion of participants with inflammation reduction as assessed on an Investigator Inflammation Assessment (IIA) Score | Up to Week 26
  The Investigator assesses the inflammation status of the target ulcer at the specified visits according to the scales.
Mean time to occurrence of a new PG ulcer(s) | Up to Week 52
  Mean time to occurrence of a new PG ulcer(s) is assessed.
Mean time to healing of target ulcer | Up to Week 52
  The PG Area Reduction (PGAR) is calculated as the percentage area change in the target PG ulcer from Baseline.
Proportion of participants achieving healing per PGAR for the target ulcer | Week 52
  The PG Area Reduction (PGAR) is calculated as the percentage area change in the target PG ulcer from Baseline.
Proportion of participants who have achieved target PGAR | Up to Week 26
  The PG Area Reduction (PGAR) is calculated as the percentage area change in the target PG ulcer from Baseline.
Percentage change in target Pyoderma Gangrenosum (PG) ulcer area | Up to Week 26
  The percentage change in target PG ulcer area is assessed.
Proportion of participants achieving PGA 0 | Week 6 and Week 26
  The Investigator assesses the global improvement of all ulcers including the target ulcer according to the scales at the specified visits.
Change from Baseline in Pain as measured by Numerical Rating Scale (NRS) | Week 6 and Week 26
  The Numerical Rating Scale of Pain sheet will be filled out in the office by participants at the designated visits.
Changes from baseline in the proportion of participants taking analgesics | Week 6 and Week 26
  Proportion of participants taking analgesics is assessed.
Velocities of healing | Up to Week 26
  This is assessed from baseline.
Proportion of participants achieving ulcer healing as assessed by PGAR | Week 6
  The PG Area Reduction (PGAR) is calculated as the percentage area change in the target PG ulcer from Baseline.
Proportion of participants achieving PGA 0 of all PG ulcers | Week 52
  The Investigator assesses the global improvement of all ulcers including the target ulcer according to the scales at the specified visits.
Mean time to relapse of the target PG ulcer | Up to Week 26
  The PG Area Reduction (PGAR) is calculated as the percentage area change in the target PG ulcer from Baseline.
Mean time to healing as defined by PGAR | Up to Week 26
  The PG Area Reduction (PGAR) is calculated as the percentage area change in the target PG ulcer from Baseline.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (20):
- Japan (20):
  - Nagoya City University Hospital /ID# 164510, Nagoya, Aichi-ken
  - Juntendo University Urayasu Hospital /ID# 164422, Urayasu Shi, Chiba
  - Fukuoka University Hospital /ID# 164416, Fukuoka, Fukuoka
  - Fukushima Medical University Hospital /ID# 164358, Fukushima, Fukushima
  - Gunma University Hospital /ID# 164464, Maebashi, Gunma
  - Asahikawa Medical University Hospital /ID# 164589, Asahikawa-shi, Hokkaido
  - Showa University Fujigaoka Hospital /ID# 164406, Yokohama, Kanagawa
  - Mie University Hospital /ID# 164389, Tsu, Mie-ken
  - Tohoku University Hospital /ID# 164360, Sendai, Miyagi
  - Shinshu University Hospital /ID# 164852, Matsumoto-shi, Nagano
  - Nagasaki University Hospital /ID# 167604, Nagasaki, Nagasaki
  - University of the Ryukyus Hospital /ID# 164981, Nakagami-gun, Okinawa
  - Hamamatsu University Hospital /ID# 165890, Hamamatsu, Shizuoka
  - Tokushima University Hospital /ID# 164359, Tokushima, Tokushima
  - Teikyo University Hospital /ID# 165665, Itabashi-ku, Tokyo
  - Tokyo Medical University Hospital /ID# 165810, Shinjuku-ku, Tokyo
  - Keio University Hospital /ID# 165680, Shinjuku-ku, Tokyo
  - Yamaguchi University Hospital /ID# 164562, Ube-shi, Yamaguchi
  - Kansai Medical Univ Hosp /ID# 165802, Hirakata-shi, Osaka
  - Hokkaido University Hospital /ID# 164419, Sapporo

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/clinical-trials/adalimumab_M16-119.pdf